CLINICAL TRIAL: NCT03697031
Title: The Impact of Frozen - Thawed Blastocyst Morphological Development and Blastocoele Re-expansion on Clinical Pregnancy Outcome After One Controlled Ovarian Stimulation Cycle Using REKOVELLE®
Brief Title: Impact of Blastocyst Morphological Development and Blastocoele Re-expansion on Pregnancy Outcome After Using REKOVELLE®
Status: Terminated | Type: Observational
Why Stopped: Permanently terminated due to halt of recruitment due to COVID-19 pandemic
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000317
Record Dates: First submitted 2018-09-14; First posted 2018-10-05 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2021-10

CONDITIONS: Controlled Ovarian Stimulation
MeSH Terms: interventions — follitropin delta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- REKOVELLE®: Follitropin Delta
  Interventions: Drug: Follitropin Delta

INTERVENTIONS:
Drug: Follitropin Delta — The Intervention (solution for injection) is delivered with an injection pen. For women with AMH <15 pmol/L the daily dose is 12 micrograms, irrespective of body weight. For women with AMH ≥15 pmol/L the daily dose decreases from 0.19 to 0.10 micrograms/kg by increasing AMH concentration. The maximum daily dose for the first treatment cycle is 12 micrograms.
  For subsequent treatment cycles, the daily dose of REKOVELLE® should be maintained or modified according to the patient's ovarian response in the previous cycle. Based on the ovarian hypo/hyper-response in the previous cycle, the daily dose in the subsequent cycle should be increased (by 25% or 50%) or decreased (by 20% or 33%). The maximum daily dose is 24 micrograms.

SUMMARY:
The purpose of this observational study is to examine the development and appearance of embryos before and after freezing following a single controlled ovarian stimulation cycle using REKOVELLE® (follitropin delta) as the recombinant follicular stimulating hormone (rFSH) for controlled ovarian stimulation. The primary objective of the study is to examine how specific factors of embryo development or appearance are related to the chance of becoming pregnant.

The ovarian stimulation protocol with REKOVELLE®, a new rFSH prescribed for ovarian stimulation, is individualised with a dosing regimen that is based on two parameters: the body weight and the level of a hormone, the anti-Müllerian hormone, (AMH), a parameter used to predict how the ovaries will respond to the ovarian stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective single embryo transfer (e-SET) in a frozen embryo replacement (FER) treatment where the frozen blastocyst was obtained from an IVF or intracytoplasmic sperm injection (ICSI) cycle following controlled ovarian stimulation with REKOVELLE® .
* Women are prescribed REKOVELLE® for their IVF or ICSI according to the approved label.
* Morphological measurements and clinical outcomes are available for the fresh embryos obtained from the IVF or ICSI cycle.
* Willing and able to understand Danish or English patient information.
* Willingness and ability to provide written informed consent.

Exclusion Criteria:

* Patients with any contraindication for treatment with REKOVELLE® for controlled ovarian stimulation.
* Patients with contraindication for undergoing assisted reproductive technologies (ART) such as an IVF or ICSI cycle.
* Oocyte donors.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: The study aims to enroll between 1200 and 1500 cycles which is estimated to be sufficient for observing 616 single frozen-thawed blastocyst transfers. Patients can contribute data from one or more frozen-thawed blastocyst transfers. Further, the patient cohort will be recruited among the patient population of 8-10 public and private in vitro fertilization (IVF) clinics in Denmark.
Sampling Method: Probability Sample
Enrollment: 362 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 7 weeks after each embryo transfer
  Clinical pregnancy is defined as at least one intrauterine gestational sac with fetal heart beat at week 7, from frozen thawed blastocysts. The correlation between morphological parameters (blastocyst score, timelapse score, blastocoele re-expansion) and clinical pregnancy rate will be assessed.

SECONDARY OUTCOMES:
Cumulative clinical pregnancy rate | Up to 24 months
  The cumulative clinical pregnancy rate will be calculated based on all participants included in the study and all clinical pregnancies recorded from fresh and frozen-thawed blastocyst transfers as the fraction of participants with at least one positive clinical pregnancy. The cumulative pregnancy rate will be plotted versus transfer number and versus time from start of REKOVELLE® treatment.
Positive βhCG result (blood or urinary pregnancy test) | Up to 24 months
Use of the algorithm-based individualized dosing regimen with REKOVELLE® | At the day of the consultation visit where the daily dose of REKOVELLE® is decided
  Use of the Ferring developed dosing app for the daily dose calculation. The daily dose is calculated with body weight in kilograms or pounds and AMH serum level in pmoL/L or ng/ml to define the daily dose of REKOVELLE® in micrograms.
Daily dose of REKOVELLE® administered | From day 1 up to day 20 of REKOVELLE® stimulation
  Daily dose of REKOVELLE® in micrograms is recorded.
Number of days of treatment with REKOVELLE® | From day 1 up to day 20 of REKOVELLE® stimulation
Day of REKOVELLE® stimulation start | At the day of the first REKOVELLE® injection during the ovarian stimulation treatment
  The time point of the start of the stimulation is decided at the discretion of the investigator.
Day of REKOVELLE® stimulation end | At the day of the last REKOVELLE® injection during the ovarian stimulation treatment
  The time point of the end of the stimulation is decided at the discretion of the investigator.
Any deviation in REKOVELLE® administration | From day 1 up to day 20 of REKOVELLE® stimulation
  REKOVELLE® should be used according to the approved label, any possible deviations such as different starting dose or dose adjustment during stimulation will be recorded and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (1):
- Ciconia, VivaNeo (there may be other sites in this country), Højbjerg, Denmark

REFERENCES:
- [Result] Gabrielsen A, Iversen LH, Fedder J, Eskildsen TV, Englund AL, Hansen SR, Pinton P. Pre-Vitrification and Post-Warming Variables of Vitrified-Warmed Blastocysts That Are Predictable for Implantation. J Clin Med. 2023 Oct 6;12(19):6389. doi: 10.3390/jcm12196389. PMID 37835035